CLINICAL TRIAL: NCT04603430
Title: The Impact of the STEPS Program: A Qualitative Study
Status: Completed | Type: Observational
Sponsor: Utica College (Other)
Responsible Party: Principal Investigator, Gabriele Moriello, Associate Professor, Utica College
Other Study IDs: 827
Record Dates: First submitted 2020-06-16; First posted 2020-10-26 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Health Promotion
Keywords: physical therapy students; health promotion; seniors; learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physical Therapy Students: Students will be participating in a focus group and completing a survey.
  Interventions: Other: Participation in a community wellness program
- Senior STEPS Participants: Seniors will be participating in a focus group, completing a survey, and researchers will be conducting a retrospective chart review on relevant documented health outcomes of the STEPS program.
  Interventions: Other: Participation in a community wellness program

INTERVENTIONS:
Other: Participation in a community wellness program — Participation in the STEPS program, a physical therapy student-run community wellness program for local seniors.

SUMMARY:
The STEPS program is a wellness program where senior citizens are partnered with Doctor of Physical Therapy (DPT) students, who design individualized fitness plans for each senior participant. In both the Spring and Fall semesters, first- and second year DPT student teams provide guided interventions based upon the fitness goals and initial examination findings of each participant. Program sessions are held once a week for one hour at a local senior wellness center located in Utica, NY. Facility membership requirements include a small annual membership fee and stipulate that members must be 55 years of age or older. The STEPS participants are recruited primarily by word of mouth.

The aim of the STEPS program is to provide an accessible fitness service to improve the health of the Utica community while also supplementing the clinical experiences of students enrolled in the DPT program at Utica College. The program gives students an opportunity to practice clinical skills and reasoning on a weekly basis, and establishes a mentorship component between students. Second-year students are enrolled in a clinical education course for both the Fall (DPT 689) and Spring semesters (DPT 699). Examination and interventions are documented on the WebPT electronic medical record system. Participant reassessments are conducted twice, halfway through the semester and again at the end of the program.

PURPOSE OF STUDY Clinics and health programs facilitated by students allow clinical experiences to be interwoven throughout the curriculum and provide students with the opportunity to learn and serve in their community. Research regarding these programs has primarily centered around pro-bono clinics run by medical students, and has been limited to the impact these programs have upon learning. No research has been conducted regarding how a local senior wellness program, such as the STEPS program, impacts senior fitness and DPT student engagement. This study will assess the effect that the STEPS program has upon the health of local seniors, while also qualitatively investigating the impact that the program has had upon the lives of local seniors and students.

In order to answer these research questions, a retrospective chart review will be conducted to evaluate the functional outcomes of participating seniors. Additionally, qualitative focus groups will be convened to reflect upon the impact that the STEPS program has had upon the seniors and students.

DETAILED DESCRIPTION:
STUDY DESIGN A mixed-method study design will be used to assess functional outcomes of the Students Teaching Elderly Prevention and Safety (STEPS) program on senior participants, as well as the impact of the program on both participants and students. In order to assess functional outcomes, a retrospective chart review will be conducted on a convenience sample of participants enrolled in the STEPS program from September 2018 to April 2019.

In order to explore participant and student perspectives of the STEPS program, a Glaserian grounded theory approach will be utilized. Grounded theory is a qualitative research methodology commonly employed in healthcare research due to its inductive, systematic process of gathering and interpreting data. Data gleaned from focus groups is continuously analyzed for patterns, from which a thematic consensus emerges. Semi -structured interview questions will be proposed to focus groups of students and senior participants who were involved in the STEPS program during the study time frame. Prior to starting the focus group discussion, subjects will be given a demographic survey to complete.

DEMOGRAPHIC SURVEYS Demographic information will be collected from senior participants and students via a written survey filled out prior to the focus group session.

INTERVIEW QUESTIONS Questions will be pilot tested with a purposive sample of eligible STEPS participants and students. Questions will be used to direct the focus groups, however, focus group discussion will be not restricted to these topics, as the Glaserian grounded theory approach allows for focus group members to guide the discussion process. Depending on feedback gained from pilot focus group sessions, questions may be modified.

PILOT INTERVIEWS In order to assess the construct validity of proposed focus group questions, prospective questions will be pilot tested with a group of seniors and students who participated in the STEPS program prior to the 2018-2019 academic year. Focus groups of pilot testers will be conducted in a manner similar to their respective demographic cohort. Focus groups of student pilot testers will be convened over a private virtual chat platform. Focus groups of senior pilot testers will be convened in a private virtual chat room. Each pilot sessions will last for fort-five to sixty-minutes, and will end when saturation is achieved. One or two researchers will facilitate the focus groups and another researcher will observe the session.

STEPS PARTICIPANT INTERVIEWS In order to assess the impact that the STEPS program has upon seniors, focus groups of 4 to 6 subjects will be convened for forty-five to sixty-minute-long sessions in a private virtual chat room. Sessions will end when saturation is met, meaning that no new insights are being revealed by focus group members. One or two researchers will facilitate the focus groups and another researcher will observe the focus group and take field notes. All researchers will receive training regarding proctoring focus groups. Focus groups will be conducted between June 2020 and November 2020 and will be audio-taped and later transcribed by the researchers. After transcription is complete, transcripts will be reviewed by research participants to confirm that transcription and initial interpretation objectively captured participant insights.

STUDENT INTERVIEWS In order to assess the impact that the STEPS program has upon students, focus groups of 4 to 6 subjects will be convened for forty-five to sixty-minute-long sessions in a private virtual chat platform. Sessions will end when saturation is met, meaning that no new insights are being revealed by focus group members. One or two researchers will facilitate the focus groups and another researcher will observe the focus group and take field notes. The focus group facilitators have had no prior relationship with student participants. No-one else, aside from focus group members and researchers, will be present during the sessions. Focus groups will be conducted between June 2020 and November 2020 and will be audio-taped and later transcribed by the researchers. After transcription is complete, transcripts will be reviewed by research participants to confirm that transcription and initial interpretation objectively captured participant insights.

ELIGIBILITY:
Inclusion Criteria:

Participated in the STEPS program during the 2018-2019 academic year as either a senior participant or a physical therapy student from the Class of 2020.

Exclusion Criteria:

Did no participate in the STEPS program during the 2018-2019 academic year as either a senior participant or a physical therapy student from the Class of 2020.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participated in the STEPS program during the 2018-2019 academic year as either a senior participant or a physical therapy student from the Class of 2020.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Psychosocial impact of the STEPS program on seniors and students | 1 year
  Using qualitative data collected from focus groups to determine how the program impacted physical therapy students and seniors.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Moriello, PT, PhD, Study Director — Utica College
Locations (1):
- Utica College, Utica, New York, United States

IPD SHARING:
Plan to Share IPD: No